CLINICAL TRIAL: NCT02287389
Title: Prospective, Randomized, Open, Controlled, Multicenter Stucy of Interventional Pulmonologic Treatment of Benign Central Airway Fibrotic Stricture
Brief Title: Study of Interventional Pulmonologic Treatment of Benign Central Airway Fibrotic Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: Changhai Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Xinqiao Hospital of Chongqing (Other); China Meitan General Hospital (Other); Micro-Tech (Nanjing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAO-NO.201402024-benign; NO.201402024 (Other Grant/Funding Number: Special Fund for Scientific Research in the Public Welfare)
Record Dates: First submitted 2014-10-26; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Obstructive Airway Disease
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Cryotherapy; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- balloon dilation (Experimental): give the cases balloon dilation as the intervention
  Interventions: Device: balloon dilation
- balloon dilation plus cryotherapy (Experimental): give the cases balloon dilation plus cryotherapy as the intervention
  Interventions: Device: balloon dilation; Procedure: cryotherapy
- BD plus spiculiform electrosurgery (Experimental): give the cases balloon dilation plus spiculiform electrosurgery as the intervention
  Interventions: Device: balloon dilation; Procedure: spiculiform electrosurgery
- BD plus mitomycin C (Experimental): give the cases Balloon dilation plus mitomycin C as the intervention
  Interventions: Device: balloon dilation; Drug: mitomycin C

INTERVENTIONS:
Device: balloon dilation
Procedure: cryotherapy
  Arms: balloon dilation plus cryotherapy
Procedure: spiculiform electrosurgery
  Arms: BD plus spiculiform electrosurgery
Drug: mitomycin C
  Arms: BD plus mitomycin C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of four interventional pulmonology techniques for the treatment of fibrotic central airway stricture.

The four techniques are：

* balloon dilation
* balloon dilation plus cryotherapy
* balloon dilation plus spiculiform electrosurgery
* balloon dilation plus mitomycin C injection

ELIGIBILITY:
Inclusion Criteria:

* tracheal incision,intubation or bronchial tuberculosis caused central airway fibrotic stenosis
* the degree of stenosis is above 50%
* estimated survival duration is longer than 3 months
* recieved no treatment one month before
* can understand the statement informed consent
* agree to enroll in the study

Exclusion Criteria:

* older than 70 years or younger than 18 years
* not fibrotic stenosis
* not central airway stenosis
* existence of lumina collapse or twisting
* severe arrhythmia, myocardial ischemia or hypertensive crisis
* coagulation disorders
* existence of severe organ disfunction
* allergic to anesthesia drugs
* refuse to participate the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
percentage of the cases that got Ⅰand Ⅱlevel remission | 3 months

SECONDARY OUTCOMES:
the values of dispnea index | 3 months
Karnofsky Physical scales | 3 months

OTHER OUTCOMES:
adverse event during the treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Faguang Jin, PhD, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China